CLINICAL TRIAL: NCT01649804
Title: A MULTICENTER, OPEN-LABEL, SINGLE ARM, LONG-TERM EXTENSION STUDY OF WA19926 TO DESCRIBE SAFETY DURING TREATMENT WITH TOCILIZUMAB IN PATIENTS WITH EARLY, MODERATE TO SEVERE RHEUMATOID ARTHRITIS
Brief Title: A Long-Term Safety Extension Study of WA19926 in Participants With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28146; 2011-006125-14 (EudraCT Number)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Results first posted 2016-09-22 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- RoActemra/Actemra single arm (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg intravenously every 4 weeks for 104 weeks

SUMMARY:
This extension study of WA19926 will assess the long-term safety and the efficacy of RoActemra/Actemra (tocilizumab) treatment in participants with rheumatoid arthritis. Participants who have completed the core study WA19926 are eligible to participate. Participants will receive RoActemra/Actemra 8 mg/kg intravenously every 4 weeks. The anticipated time on study drug is 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/=18 years of age who have completed the core study WA19926 and according to the investigator may benefit from RoActemra/Actemra treatment
* No current or recent adverse event or laboratory finding preventing the use of the study drug dose at baseline
* Receiving treatment on an outpatient basis

Exclusion Criteria:

* Females who are pregnant
* Participants who have prematurely withdrawn from the core study WA19926 for any reason
* Treatment with any investigational drug since the last administration of the study drug in the core study WA19926
* Treatment with an anti-tumor necrosis (TNF), anti-interleukin 1 agent or T-cell costimulation modulator since the last administration of the study drug in the core study WA19926
* Immunization with live/attenuated vaccine since the last administration of the study drug in the core study WA19926
* Diagnosis since the last WA19926 visit of rheumatic autoimmune disease or inflammatory joint disease other than rheumatoid arthritis
* Abnormal laboratory values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Hungary (3):
  - Budapest
  - Debrecen
  - Eger

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Tocilizumab (RoActemra/Actemra) 8 milligram/kilogram (mg/kg) intravenously every 4 weeks for 104 weeks. Dose could be reduced due to safety reasons at any time during the study.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 12
Completed | 4
Not Completed | 8
Not completed — Administrative/Other | 8

BASELINE CHARACTERISTICS:
Population: Analysis population included all the enrolled participants in the study.
Groups:
- Tocilizumab: Tocilizumab (RoActemra/Actemra) 8 mg/kg intravenously every 4 weeks for 104 weeks. Dose could be reduced due to safety reasons at any time during the study.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.25 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs of Special Interest (AESIs)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. A SAE was any experience that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant. Adverse Events of Special Interest for this study were: Serious and/or medically significant infections; myocardial infarction/Acute coronary syndrome; Gastrointestinal perforation; Malignancies; Anaphylaxis/hypersensitivity reactions; Demyelinating disorders; Stroke and Serious and/or medically significant bleeding and hepatic events.
Time Frame: End of Study (Week 104 or early withdrawal)
Population: Analysis population included all the enrolled participants in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 12
percentage of participants
  AEs | 75
  SAEs | 0
  AESI | 0

2. Secondary Outcome: Number of Participants With Remission, Low, Medium, and High Disease Activity, as Measured by Disease Activity Index 28 Erythrocyte Sedimentation Rate (DAS28-ESR)
Description: The DAS28 (ESR) score is a measure of the participant's disease activity. It is calculated using the tender joint count (28 joints), swollen joint count (28 joints), erythrocyte sedimentation rate (ESR) and general health status. The DAS28-ESR scale ranges from 0 to 10, where higher scores represent higher disease activity. DAS28 <=3.2 implied low disease activity, DAS >3.2 to 5.1 implied moderate disease activity, DAS >5.1 implied high disease activity, and DAS28 <2.6 = clinical remission.
Time Frame: Screening and End of Study (Week 104 or early withdrawal)
Population: Analysis population included all the enrolled participants in the study.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 12
participants
  Remission (Baseline) | 5
  Low Disease Activity (Baseline) | 1
  Moderate Disease Activity (Baseline) | 4
  High Disease Activity (Baseline) | 2
  Remission (End of Study) | 10
  Low Disease Activity (End of Study) | 1
  Moderate Disease Activity (End of Study) | 0
  High Disease Activity (End of Study) | 1

3. Secondary Outcome: Number of Participants With Remission, Low, Medium, and High Disease Activity, as Measured by Simplified Disease Activity Index (SDAI)
Description: The SDAI was defined as the numerical sum of 5 outcome parameters: tender and swollen joint count (based on a 28-joint assessment), participant and physician global assessment of disease activity on a 100 millimeter (mm) Visual analogue scale (VAS) (VAS; 0 = no disease activity and 100 = worst disease activity) and level of C-reactive protein (CRP) (milligram per deciliter [mg/dl], normal < 1 mg/dl). SDAI total score = 0-86 where a higher score reflects worsening disease. SDAI <=3.3 indicates clinical remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high (or severe) disease activity.
Time Frame: Screening and End of Study (Week 104 or early withdrawal)
Population: Analysis population included all the enrolled participants in the study.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 12
participants
  Remission (Baseline) | 0
  Low Disease Activity (Baseline) | 6
  Moderate Disease Activity (Baseline) | 3
  High Disease Activity (Baseline) | 3
  Remission (End of Study) | 3
  Low Disease Activity (End of Study) | 7
  Moderate Disease Activity (End of Study) | 1
  High Disease Activity (End of Study) | 1

4. Secondary Outcome: Number of Participants With Decreased, Unchanged, and Increased Tender Joint Count (TJC)
Description: Tender joint count was performed by a skilled assessor, evaluating 68 joints for tenderness.
Time Frame: Week 12 and Week 104
Population: Analysis population included all the evaluable participants for this outcome measure. "n" included all the participants analyzed on that particular time point.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
participants
  Decreased (Week 12; n=11) | 5
  Unchanged (Week 12; n=11) | 4
  Increased (Week 12;n=11) | 2
  Decreased (Week 104;n=4) | 2
  Unchanged (Week 104;n=4) | 2
  Increased (Week 104;n=4) | 0

5. Secondary Outcome: Number of Participants With Decreased, Unchanged, and Increased Swollen Joint Count (SJC)
Description: Swollen joint count was performed by a skilled assessor, evaluating 66 joints for swelling.
Time Frame: Week 12 and Week 104
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
participants
  Decreased (Week 12; n=11) | 3
  Unchanged (Week 12; n=11) | 7
  Increased (Week 12;n=11) | 1
  Decreased (Week 104;n=4) | 2
  Unchanged (Week 104;n=4) | 2
  Increased (Week 104;n=4) | 0

6. Secondary Outcome: Time to Rheumatoid Arthritis (RA) Flare
Description: RA flare was defined as any worsening of the participant's disease activity that in the opinion of the Investigator required treatment intensification beyond supportive therapy which included restarting of the study drug treatment. Time to RA flare was defined as the period of drug-free remission until documentation of RA flare. Drug-free remission was defined as clinical remission (based on DAS28-ESR < 2.6 and /or SDAI ≤ 3.3) for two consecutive assessment visits, followed by discontinuation of tocilizumab, at the Investigator's discretion, at the second assessment visit.
Time Frame: End of Study (Week 104 or early withdrawal)
Population: This outcome could not be evaluated as there were no participants who had achieved drug-free remission, per protocol definition.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Decreased, Unchanged, and Increased Participants Global Assessment of Disease Activity
Description: The participant global assessment of disease activity was measured using a 100 mm VAS ranging from 0=very good to 100=very bad.
Time Frame: Week 12 and Week 104
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
participants
  Decreased (Week 12; n=11) | 6
  Unchanged (Week 12; n=11) | 0
  Increased (Week 12;n=11) | 5
  Decreased (Week 104;n=4) | 2
  Unchanged (Week 104;n=4) | 0
  Increased (Week 104;n=4) | 2

8. Secondary Outcome: Number of Participants With Decreased, Unchanged, and Increased Participant Global Assessment of Pain
Description: A participant's overall assessment of pain on a VAS was assessed with a question concerning the amount of pain due to arthritis. Pain was assessed on a 100 mm VAS scale with a left-hand marker "no pain" (0 mm) or right-hand marker "extreme pain" (100 mm).
Time Frame: Week 12 and Week 104
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
participants
  Decreased (Week 12; n=11) | 7
  Unchanged (Week 12; n=11) | 4
  Increased (Week 12;n=11) | 0
  Decreased (Week 104;n=4) | 2
  Unchanged (Week 104;n=4) | 0
  Increased (Week 104;n=4) | 2

9. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The Health Assessment Questionnaire Disability Index (HAQ-DI) is a participant-completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Each item was scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores divided by the number of domains answered. Total possible scores range from 0 to 3, where 0=least difficulty, and 3=extreme difficulty.
Time Frame: End of Study (Week 104 or early withdrawal)
Population: Analysis population included all the enrolled participants in the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 12
units on a scale | 1.18 (0.953)

ADVERSE EVENTS:
Time Frame: End of Study (Week 104 or early withdrawal)
Description: An AE was any untoward medical occurrence in a study participant administered a pharmaceutical product, and which did not necessarily have a causal relationship with the treatment.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=12)
Diarrhoea (Gastrointestinal disorders) | 2
Ranula (Gastrointestinal disorders) | 1
Cystitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
White blood cell count decreased (Investigations) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Sciatica (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.